CLINICAL TRIAL: NCT06338904
Title: Efficacy of a Brief Poblem-solving Based Psychological Intervention Implemented in Different Formats for the Indicated Prevention of Suicide in Adults Over 50
Brief Title: Brief Problem-solving Intervention in Different Formats for the Prevention of Suicide in Adults Over 50
Acronym: SOLPROSU50+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, Fernando Lino Vázquez González, Full Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PID2022-141225OB-I00
Record Dates: First submitted 2024-03-02; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Suicide
Keywords: randomized controlled trial; prevention; problem solving; conference call; App; Adults over 50
MeSH Terms: conditions — Suicide; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Problem-solving-based psychological intervention delivered in a face-to-face format (PSPI-FF) (Experimental): Participants in this group will receive a problem-solving intervention for suicide prevention in a face-to-face format. The intervention will consist of 6 sessions, approximately 90 minutes in duration each, once a week, in a group format, in person.
  Interventions: Behavioral: Problem-solving-based psychological intervention
- Problem-solving-based psychological intervention delivered via telephone conference call (PSPI-CC) (Experimental): Participants in this group will receive the intervention described in a teleconference call format, with the same duration, contents, and structure.
  Interventions: Behavioral: Problem-solving-based psychological intervention
- Problem-solving-based psychological intervention delivered via a smartphone app (PSPI-A) (Experimental): Participants in this group will receive the intervention described adapted to be administered through a smartphone app, with equivalent duration, content, and structure (approximately 90 minutes to complete each of the 6 modules).
  Interventions: Behavioral: Problem-solving-based psychological intervention
- Usual care (UCCG) (No Intervention): Participants in this group will receive usual care. Usual treatment will include individual and group psychotherapy and/or psychiatric medication as determined by the health professionals they are currently consulting, whether in public or private facilities.

INTERVENTIONS:
Behavioral: Problem-solving-based psychological intervention — The intervention will include training in the components of the problem-solving model and other behavioral and cognitive skills such as detecting warning signals, monitoring mood, relaxation techniques, self-reinforcement, strategies for acting in crisis situations, engaging in enjoyable activities, mindfulness meditation techniques, or strategies for reframing irrational thoughts. It will be developed from the problem-solving model (D'Zurilla and Nezu, 1982) and will reference the indicated prevention program for depression (Vázquez et al., 2015), which has shown efficacy in reducing depressive symptoms and preventing the onset of depression episodes (Otero et al., 2015; Vázquez et al., 2013), with results on symptomatology maintained at 8 years (López et al., 2020); and the indicated prevention intervention that demonstrated efficacy in reducing suicide risk (Xavier et al., 2019).
  Arms: Problem-solving-based psychological intervention delivered in a face-to-face format (PSPI-FF); Problem-solving-based psychological intervention delivered via a smartphone app (PSPI-A); Problem-solving-based psychological intervention delivered via telephone conference call (PSPI-CC)

SUMMARY:
Suicide represents a personal tragedy and an enormous global public health problem. One of the most vulnerable groups is adults 50 years and older. Despite this stage of life is particularly amenable to the implementation of targeted suicide prevention strategies, we have few studies of the efficacy of psychological interventions, those that do exist have methodological limitations, and none were implemented in formats other than face-to-face, which limits their accessibility. There is a need for brief psychological interventions that can be administered in both face-to-face and remote formats, do not require long training periods, and are effective in different contexts: for example, problem-solving therapy. The main objective of this project is to evaluate the efficacy of a brief problem-solving psychological intervention for targeted suicide prevention in people aged 50 years and older, administered in face-to-face, conference call, and smartphone app formats. A randomized controlled trial will be performed. Participants will be recruited through healthcare centers in the Autonomous Community of Galicia (Spain). To be included, participants must: (a) be at least 50 years old, (b) reside in Galicia, and (c) present suicidal ideation. Subjects will be excluded if they: (a) present serious mental health or medical disorders; (b) have begun receiving psychological or psychopharmacological treatment in the previous two months or are participating in other suicide prevention research; (c) do not have an appropriate mobile device or sufficient fluency to communicate in Spanish, or have problems that make it impossible to participate; or (d) plan to move in the next 18 months. At pre-intervention information will be collected on sociodemographic, family, personal history, current suicide risk and other clinical variables. 212 participants will be randomly assigned to (1) a problem-solving-based psychological intervention delivered face-to-face (PSPI-FF; experimental group 1); (2) a problem-solving-based psychological intervention delivered via telephone conference call (PSPI-CC; experimental group 2); (3) a problem-solving-based psychological intervention delivered via a smartphone app (PSPI-A; experimental group 3); or (4) a usual care control group (UCCG). Participants in the experimental groups will complete the six sessions/modules of the interventions. Finally, subjects in all groups will be evaluated at post-intervention and 3, 6 and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 50 years old
* Reside in Galicia
* Present suicidal ideation

Exclusion Criteria:

* Present serious mental health or medical disorders
* Have begun receiving psychological or psychopharmacological treatment in the previous two months or are participating in other suicide prevention research
* Do not have an appropriate mobile device or sufficient fluency to communicate in Spanish, or have problems that make it impossible to participate
* Plan to move in the next 18 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline suicidal ideation to post-treatment (7 weeks), and follow-ups at 6 and 12 months. | Pre- and post-intervention (7 weeks) with follow-ups at 3, 6 and 12 months
  Suicidal ideation will be assessed using the Suicidal Ideation Scale (SSI; Beck et al., 1979), a semi-structured scale of 19 items with an internal consistency (Kuder-Richardson coefficient [KR-20]) of .89 and an inter-rater reliability (k) of .83.
Change from baseline suicidal ideation to post-treatment (7 weeks), and follow-ups at 6 and 12 months. | Pre- and post-intervention (7 weeks) with follow-ups at 3, 6 and 12 months
  Aditionally, the severity of ideation and suicidal behavior over the last month will be assessed using the Columbia Scale for assessing suicide risk (C-SSRS; Posner et al., 2011). It consists of a semi-structured interview with good convergent and discriminant validity and high sensitivity (100.0%) and specificity (99.4%) for the classification of suicidal behavior; the ideation intensity subscale showed a Cronbach's alpha of .73-.95.

SECONDARY OUTCOMES:
Change from baseline hopelessness to post-treatment (7 weeks), and follow-ups at 6 and 12 months | Pre- and post-intervention (7 weeks) with follow-ups at 3, 6 and 12 months
  Hopelessness will be assessed with the Beck Hopelessness Scale (HS; Beck et al., 1974), a self-administered instrument of 20 items with a range from 0 to 20. Higher scores mean higher hopelessness. It has an internal consistency (Kuder-Richardson 20 [KR-20]) of .93.
Change from baseline anxiety and depressive symptoms to post-treatment (7 weeks), and follow-ups at 6 and 12 months | Pre- and post-intervention (7 weeks) with follow-ups at 3, 6 and 12 months
  Anxiety and depression symptoms will be assessed with the General Health Questionnaire (GHQ-12; Goldberg & Williams, 1988), a self-administered questionnaire of 12 items designed to screen for non-psychotic psychiatric morbidity, with a range from 0 to 12. Higher scores mean higher anxiety and depressive symptoms. Its internal consistency (Cronbach's alpha) is .86 for individuals under 65 years of age and .90 for individuals aged 65 years or older.
Change from baseline reasons for living to post-treatment (7 weeks), and follow-ups at 6 and 12 months | Pre- and post-intervention (7 weeks) with follow-ups at 3, 6 and 12 months
  Deterrent reasons for attempting suicide will be assessed through the Reasons for Living Inventory (RFL; Linehan et al., 1983), a self-administered instrument of 48 items across six subscales, with a range from 48 to 288. Higher scores mean that individuals exhibit higher reasons for living. Internal consistencies (Cronbach's alphas) range from .72 to .89.
Change from baseline impulsivity to post-treatment (7 weeks), and follow-ups at 6 and 12 months | Pre- and post-intervention (7 weeks) with follow-ups at 3, 6 and 12 months
  Impulsivity will be assessed using the Barratt Impulsiveness Scale (BIS-11; Patton et al., 1995), a self-administered instrument of 30 items, with a range from 30 to 120. Higher scores mean higher impulsivity. Its internal consistencies (Cronbach's alphas) range from .79 to .82.
Change from baseline problem-solving skills to post-treatment (7 weeks), and follow-ups at 6 and 12 months | Pre- and post-intervention (7 weeks) with follow-ups at 3, 6 and 12 months
  Problem-solving skills will be assessed with the Revised Social Problem-Solving Inventory (SPSI-R; D'Zurilla et al., 1997), an inventory of 52 items with a range from 0 to 208, and an internal consistency (Cronbach's alpha) ranging from .68 to .92.
Change from baseline social support to post-treatment (7 weeks), and follow-ups at 6 and 12 months | Pre- and post-intervention (7 weeks) with follow-ups at 3, 6 and 12 months
  Social support will be evaluated with the DUKE-UNC Functional Social Support Questionnaire (Duke-UNC-11; Broadhead et al., 1988), an 11-item questionnaire with a range from 11 to 55 and an internal consistency (Cronbach's alpha) of .90. Higher scores mean higher social support.
Change from baseline syndrome of clinical anger to post-treatment (7 weeks), and follow-ups at 6 and 12 months | Pre- and post-intervention (7 weeks) with follow-ups at 3, 6 and 12 months
  The anger syndrome will be assessed with the Clinical Anger Scale (CAS; Snell et al., 1995), a self-administered instrument of 21 items with a range from 0 to 63, and an internal consistency (Cronbach's alpha) of .94. Higher scores correspond to greater clinical anger.
Treatment adherence | During the intervention sessions (6 weeks)]
  Treatment adherence will be assessed by recording the number of sessions attended or modules completed by each participant, and the number of intersession tasks completed.
Satisfaction with the service received | Post-intervention (7 weeks)
  Satisfaction with the intervention will be evaluated using the Client Satisfaction Questionnaire (CSQ-8; Larsen et al., 1979), an 8-item scale whose total score varies from 8 to 32, where a higher score indicates greater satisfaction with the service received. It has an internal consistency (Cronbach's alpha) of .80.

OTHER OUTCOMES:
Sociodemographic, familial, personal history, and current suicide risk variables | Pre-intervention.
  These variables will be assessed using a hetero-administered questionnaire, developed ad hoc for this study, following the recommended criteria in the Clinical Practice Guideline for the Prevention and Treatment of Suicidal Behavior (Grupo de Trabajo de la Guía de Práctica Clínica de Prevención y Tratamiento de la Conducta Suicida, 2012/2020). This questionnaire will include information on: sex, age, marital status, living arrangements, rural/urban setting, education level, main activity, family monthly income, characteristics of suicidal ideation (e.g., potential plans, access to lethal means, intent to die, previous suicide attempts); present/past risk factors (e.g., risk factors related to psychological and psychiatric problems, family history of suicidal behavior and mental disorder, history of physical abuse or sexual abuse); and health and psychosocial stress factors (e.g., presence of chronic illness, financial problems).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L. Vazquez González, PhD., Principal Investigator — University of Santiago de Compostela; Ángela J. Torres Iglesias, PhD., Principal Investigator — University of Santiago de Compostela
Locations (1):
- Research Group on Mental Health and Psychopatology, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Zurilla TJ, Nezu, A. Social problem solving in adults. In: Kendall PC (editor). Advances in cognitive-behavioral research on therapy. New York: Academic Press; 1982. vol. 1, p. 202-74.
- [Background] Vázquez FL, Otero P, Blanco V, Torres AJ. Terapia de solución de problemas para la depresión: una breve guía práctica en grupo. Madrid: Alianza Editorial. 2015.
- [Background] Otero P, Smit F, Cuijpers P, Torres A, Blanco V, Vazquez FL. Long-term efficacy of indicated prevention of depression in non-professional caregivers: randomized controlled trial. Psychol Med. 2015 May;45(7):1401-12. doi: 10.1017/S0033291714002505. Epub 2014 Oct 21. PMID 25331992
- [Background] Vazquez Gonzalez FL, Otero Otero P, Torres Iglesias A, Hermida Garcia E, Blanco Seoane V, Diaz Fernandez O. A brief problem-solving indicated-prevention intervention for prevention of depression in nonprofessional caregivers. Psicothema. 2013 Feb;25(1):87-92. doi: 10.7334/psicothema2012.89. PMID 23336549
- [Background] Lopez L, Smit F, Cuijpers P, Otero P, Blanco V, Torres A, Vazquez FL. Problem-solving intervention to prevent depression in non-professional caregivers: a randomized controlled trial with 8 years of follow-up. Psychol Med. 2020 Apr;50(6):1002-1009. doi: 10.1017/S0033291719000916. Epub 2019 Apr 24. PMID 31017076
- [Background] Xavier A, Otero P, Blanco V, Vazquez FL. Efficacy of a problem-solving intervention for the indicated prevention of suicidal risk in young Brazilians: Randomized controlled trial. Suicide Life Threat Behav. 2019 Dec;49(6):1746-1761. doi: 10.1111/sltb.12568. Epub 2019 Jun 25. PMID 31237377
- [Background] Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. J Consult Clin Psychol. 1979 Apr;47(2):343-52. doi: 10.1037//0022-006x.47.2.343. No abstract available. PMID 469082
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Background] Goldberg D, Williams P.. A user's guide to the General Health Questionnaire. Windsor: NFER-Nelson. 1988.
- [Background] Linehan MM, Goodstein JL, Nielsen SL, Chiles JA. Reasons for staying alive when you are thinking of killing yourself: the reasons for living inventory. J Consult Clin Psychol. 1983 Apr;51(2):276-86. doi: 10.1037//0022-006x.51.2.276. No abstract available. PMID 6841772
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Background] D'Zurilla TJ, Nezu AM, Maydeu-Olivares A.Manual for the social problem solving inventory-revised. North Tonawanda, NY: Multi-Health Systems. 1997.
- [Background] Broadhead WE, Gehlbach SH, de Gruy FV, Kaplan BH. The Duke-UNC Functional Social Support Questionnaire. Measurement of social support in family medicine patients. Med Care. 1988 Jul;26(7):709-23. doi: 10.1097/00005650-198807000-00006. PMID 3393031
- [Background] Snell WE Jr, Gum S, Shuck RL, Mosley JA, Hite TL. The Clinical Anger Scale: preliminary reliability and validity. J Clin Psychol. 1995 Mar;51(2):215-26. doi: 10.1002/1097-4679(199503)51:23.0.co;2-z. PMID 7797645
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Grupo de Trabajo de la Guía de Práctica Clínica de Prevención y Tratamiento de la Conducta Suicida Guía de práctica clínica de prevención y tratamiento de la conducta suicida [Clinical Practice Guideline for the Prevention and Treatment of Suicidal Behavior] (Ed. Rev. 2020).Santiago de Compostela: Plan de calidad para el Sistema Nacional de Salud del Ministerio de Sanidad, Política Social e Igualdad, Agencia de Evaluación de Tecnologías Sanitarias de Galicia (avaliat-t). 2012.
- [Derived] Vazquez FL, Torres AJ, Blanco V, Bouza Q, Otero P, Andrade E, Simon MA, Bueno AM, Arrojo M, Paramo M, Fernandez A. Brief psychological intervention for suicide prevention based on problem-solving applied in different formats to people over 50 years old: protocol for a randomized controlled trial. BMC Psychiatry. 2024 Sep 27;24(1):628. doi: 10.1186/s12888-024-06076-5. PMID 39334120